CLINICAL TRIAL: NCT01626326
Title: Evaluation of a Stop Smoking iPhone App
Brief Title: San Francisco Stop Smoking App - Pilot Study
Acronym: TCapp-1
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: TCapp-1
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Recruitment
Keywords: smoking; smoking cessation; mobile app
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stop smoking app: Stop smoking iPhone research app provided at no charge via the iTunes store
  Interventions: Behavioral: San Francisco Stop Smoking iPhone app

INTERVENTIONS:
Behavioral: San Francisco Stop Smoking iPhone app — iPhone app designed to help people quit smoking

SUMMARY:
This is an initial pilot study to determine whether people will use a research version of an iPhone Stop Smoking app. The investigators primary measures will consist of rates of recruitment (that is, number of people installing the app), use of the app, and completion of follow-up surveys regarding self-reported smoking status. The investigators secondary measure will be obtained quit rates and number of cigarettes smoked before and after using the app.

To enter the study, participants must download the app from iTunes at:

https://itunes.apple.com/us/app/san-francisco-stop-smoking/id522832206?mt=8

DETAILED DESCRIPTION:
The investigators research team has developed smoking cessation self-help tools administered as printed brochures and Internet stop smoking sites. These self-help tools have demonstrated quit rates similar to those obtained with the nicotine patch. The investigators now want to see if mobile device apps might also help people quit.

This is the investigators first pilot study with a research version of the investigators stop smoking app for the iPhone. The investigators want to get estimates of how many people will download the app per month, how many will actually use the app, and how many will provide follow-up information on whether they quit, and if not, how many cigarettes they are smoking now. The investigators will use this information to plan a randomized controlled trial to determine efficacy of the app for stopping smoking.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must download the iPhone app from iTunes at: https://itunes.apple.com/us/app/san-francisco-stop-smoking/id522832206?mt=8

Exclusion Criteria:

* less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who use iPhone stop smoking apps
Sampling Method: Non-Probability Sample
Enrollment: 9935 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | Three years
  Rates of recruitment into study (defined as number of users who provide consent by installing the app)

SECONDARY OUTCOMES:
Utilization | One year
  Proportion of consented users who enter data into the app
Follow-up completion rates | One year
  Proportion of consented users who provide smoking data at follow-ups
Quit rates | 1, 3, and 6 months
  Self-reported quit rates at 1, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Muñoz, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psychiatry at San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Munoz RF, Marin BV, Posner SF, Perez-Stable EJ. Mood management mail intervention increases abstinence rates for Spanish-speaking Latino smokers. Am J Community Psychol. 1997 Jun;25(3):325-43. doi: 10.1023/a:1024676626955. PMID 9332966